CLINICAL TRIAL: NCT04378556
Title: Improving Dietary Protein Intake in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1151456-1
Record Dates: First submitted 2020-04-27; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Protein intake; Coaching; Strength

STUDY DESIGN:
Intervention Model Description: Repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition (Other): All participants received diet coaching, nutrition education and a per-meal protein prescription.
  Interventions: Behavioral: Nutritional coaching

INTERVENTIONS:
Behavioral: Nutritional coaching — Participants were provided with nutrition education and a per-meal protein prescription followed by 9 weeks of nutritional coaching.

SUMMARY:
A pilot, single-arm investigation used coaching, nutrition education, and a per-meal protein prescription to assess impact on protein intake, muscle strength and function in older adults.

DETAILED DESCRIPTION:
Objective: To evaluate the effects of nutrition education, diet coaching, and a protein prescription (PP) on protein intake, and associations with muscle strength and function. Design: Prospective pretest posttest single-arm study. Setting: Urban area, East coast of South Florida. Participants: Older adults. Intervention: 10-week telephone-based diet coaching, nutrition education and a per-meal PP. Measurements: Protein and energy intakes, weight, grip strength (GS), and 5-chair-rise (5CR), timed up and go (TUG), 3-meter walk (3mW) tests at baseline and 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 years or older,
* Community-dwelling (living independently),
* Able to provide consent,
* Able to understand and respond to questions or instructions in English,
* Have a working telephone (for coaching sessions),
* Willingness to consume protein-containing animal products
* Willingness to make changes to the diet

Exclusion Criteria:

* Self-reported information that they have been told by a medical doctor that they have kidney (renal) disease.
* Vegan dietary practices,
* Refusal to make changes to usual dietary protein intake, or a usual dietary protein intake that meets recommendations.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Protein intake | Change from baseline to 10 weeks
  Protein intake (g/kg/body weight) per day

SECONDARY OUTCOMES:
Change in Grip strength | Change from baseline to 10 weeks
  Grip strength measured using dynamometer
Change in Timed Up and Go Test | Change from baseline to 10 weeks
  The timed up and go test measures the time (in seconds) that it takes to stand up from a seated position in a chair, walk 3 meters away from the chair at a comfortable pace to a line on the floor, turn around, walk back, and sit back down in the chair.
Change in 3 meter walk | Change from baseline to 10 weeks
  The 3-meter walk test measures the time (in seconds) that it takes to stand up from a seated position in a chair and walk 3 meters away from the chair at a comfortable pace to a line on the floor
Change in 5-Chair Rise Stand Test | Change from baseline to 10 weeks
  The 5 chair rise stand test requires participants to stand up 5 times without hand assistance from a straight back chair without an armrest. The time required to complete the 5 chair rises is recorded.
Change in Short Performance Physical Battery Score | Change from baseline to 10 weeks
  The Short Physical Performance Battery (SPPB) consists of timed measures of balance, 3-meter walk, and 5-chair rises. The balance portion requires participants to stand with feet next to each other, the toes of one foot next to the heel of the other foot, and heel to toe for a 10 second duration. Scores are assigned based on the number of seconds the participant can stand in the position for balance. Scores for the chair rise and 3 meter walk are based on the time taken to complete the task. The scores are totaled to arrive at the Short Performance Physical Battery Score

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No